CLINICAL TRIAL: NCT01923454
Title: Immediate Anterior Chamber Paracentesis With A 30-Gauge Needle for Acute Primary Angle - Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK001
Record Dates: First submitted 2013-08-04; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Glaucoma, Angle-closure
Keywords: paracentesis; primary acute angle closure; iridotomy; filtration; glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure; Glaucoma | interventions — Paracentesis; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paracentesis (Experimental): Immediate anterior chamber paracentesis (ACP) with a 30-gauge needle as an initial treatment for acute primary angle closure.
  Acetamide, given in this study, is a standard treatment for acute angle-closure glaucoma. The participant will receive 1 tablet(250mg) at 1 hours after paracentesis. The following dose will be adjusted according to the level of IOP. The maximal dose is 4 tablets per day. It will be discontinued if the IOP is less than 21 mmHg.
  All affected eyes will receive laser peripheral iridotomy with 24 hours after presentation. This a standard treatment for Acute angle-closure glaucoma
  Interventions: Procedure: Paracentesis; Drug: Acetazolamide; Procedure: Peripheral iridotomy

INTERVENTIONS:
Procedure: Paracentesis — At presentation, patients received immediate anterior chamber paracentesis with a 30-gauge needle. The intraocular pressure (IOP) was recorded at immediately, 15 and 30 minutes, and then 1, 24 and 48 hours after paracentesis. The IOP was compared between before paracentesis and each time-point after paracentesis. All affected eyes received antiglaucomatous medications 60 minutes after ACP and underwent peripheral iridotomy within 24 hours.
  Other Names: A 30-gauge needle
Drug: Acetazolamide — All participants will receive oral acetazolamide (250 mg) 1 tablet at 1 hour after paracentesis to lower the intraocular pressure. After that, the dose of acetazolamide will be adjusted according to the level of intraocular pressure. If the eye pressure goes to normal (lower than 21 mmHg), acetazolamide will be discontinued.
  Other Names: Acetazolamide (Diamox 250 mg)
Procedure: Peripheral iridotomy — All affected eyes underwent laser peripheral iridotomy within 24 hours after presentation. This procedure is a standard treatment for acute angle-closure. The fellow eyes will receive laser peripheral iridotomy in the same occasion or later to prevent acute angle-closure in the future.
  Other Names: Laser peripheral iridotomy

SUMMARY:
This study was to evaluate the efficacy and safety of immediate anterior chamber paracentesis (ACP) with a 30-gauge needle as an initial treatment for acute primary angle closure (APAC).

DETAILED DESCRIPTION:
This is a prospective study from patients with APAC presenting at the Faculty of Medicine Siriraj Hospital, Bangkok, Thailand in 2005. At presentation, patients received immediate ACP with a 30-gauge needle. The IOP, best corrected visual acuity (BCVA), corneal edema grading, pupil size and symptoms were recorded at immediately, 15 and 30 minutes, and then 1, 24 and 48 hours after paracentesis. All affected eyes received antiglaucomatous medications 60 minutes after ACP and underwent peripheral iridotomy within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 year old with the first attack of APAC
* IOP of more than or equal to 40 mmHg.

Exclusion Criteria:

* patient unable to cooperate for paracentesis
* patients with APAC in the only remaining eye
* patients received any glaucoma treatments prior to the study
* patients with secondary causes of acute angle closure
* patients with intraocular inflammation or infection; (6) patients with APAC in the eye with a history of previous intraocular surgery
* patients known hypersensitive to tetracaine hydrochloride or tobramycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The Intraocular pressure (mmHg) | Change of intraocular pressure between before paracentesis and at 48 hours after paracentesis
  The intraocular pressure (IOP) was recorded at immediately(within 2 minutes after paracentesis), 15 and 30 minutes, and then 1, 24 and 48 hours after paracentesis. The change of IOP was study between before paracentesis and at each time-point. All affected eyes received antiglaucomatous medications 60 minutes after paracentesis and underwent peripheral iridotomy within 24 hours.

SECONDARY OUTCOMES:
Numbers of complications | at immediately(within 2 minutes after paracentesis), 15 and 30 minutes, and then 1, 24 and 48 hours after paracentesis.
  This is to observe the potential complications which may occur during and after paracentesis with a 30-gauge needle. Among the potential complications include lens capsular rupture, hyphema, retinal hemorrhage, hypotony and infection. The study will record each complications as numbers of events at each time-point until 48 hours after paracentesis

OTHER OUTCOMES:
visual acuity | The change of visual acuity between before paracentesisat and immediately (within 2 minutes) after paracentesis, 1 hours, 24 hours and 48 hours after paracentesis
  The study will record the visual acuity with Snellen's chart at immediately (within 2 minutes after paracentesis), 1 hours, 24 hours and 48 hours after paracentesis.

CONTACTS AND LOCATIONS:
Overall Officials: Naris Kitnarong, M.D., Principal Investigator — Mahidol University
Locations (1):
- Naris Kitnarong, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Pong JC. Anterior chamber paracentesis in patients with acute elevation of intraocular pressure. Graefes Arch Clin Exp Ophthalmol. 2008 Mar;246(3):463-4; author reply 465-6. doi: 10.1007/s00417-007-0675-5. Epub 2007 Dec 11. No abstract available. PMID 18071739
- [Result] Lam DS, Chua JK, Tham CC, Lai JS. Efficacy and safety of immediate anterior chamber paracentesis in the treatment of acute primary angle-closure glaucoma: a pilot study. Ophthalmology. 2002 Jan;109(1):64-70. doi: 10.1016/s0161-6420(01)00857-0. PMID 11772581